CLINICAL TRIAL: NCT07323758
Title: Effects of Music Application and Gum Chewing on Pain, Anxiety, and Patient Satisfaction During Episiotomy Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ayşe Sevim AKBAY KISA, Teaching Assistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 16.05.2025/155-58
Record Dates: First submitted 2025-11-14; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pain; Anxiety; Patient Satisfaction
Keywords: pain; anxiety; Patient Satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Patient Satisfaction | interventions — Music Therapy; Chewing Gum

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a three-group randomized controlled study to determine the effects of music and chewing gum on pain, anxiety, and patient satisfaction during the episiotomy repair procedure.
  Randomization The name of each group (Music Group, Chewing Gum Group, and Control Group) will be written on a piece of paper, and the group number (1, 2, and 3) will be determined by drawing lots. To ensure randomization in the study, numbers equal to the sample size (1, 2, 3, 4, 5, etc.) will be entered on the website www.random.org/ and divided into three groups, creating a random number table. The numbers in the columns determined on the website random.org/ will then be entered in the diagram below the group number determined by drawing lots. Pregnant women arriving at the delivery room and enrolled in the study will be assigned to the group they were in (Music Group, Chewing Gum Group, and Control Group) in the order they arrived.
  Intervention Group Implementation Step
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): Women in the music group will listen to their preferred music using an Music Headphones connected to speakers in the delivery room between the beginning and end of the episiotomy repair (15-20 minutes).
  Interventions: Behavioral: Music
- Gum Chewing group (Experimental): Women in the music group will listen to their preferred music using an Music Headphones connected to speakers in the delivery room between the beginning and end of the episiotomy repair (15-20 minutes).
  Gum group protocol: Women assigned to the gum group will chew plain gum between the beginning and end of the episiotomy repair (15-20 minutes). They will be asked to chew the same brand of easy-to-chew, sugar-free gum that does not contain sorbitol or xylitol. Sugar-free gum is preferred to avoid the risk of GI problems if swallowed with sorbitol-containing gum, and the risk of diarrhea if consumed in excess with xylitol. Given the risk of aspiration while chewing gum, the woman will be positioned in a semi-fowler position.
  Interventions: Behavioral: Gum Chewing
- Control group (No Intervention): Pregnant women in the control group will be administered an informed consent form, a pregnant information form, and a labor monitoring form during the active phase of the first stage. Pregnant women in the control group will not deviate from routine procedures performed in the delivery room.

INTERVENTIONS:
Behavioral: Music — No studies in the literature have investigated the use of music and chewing gum during episiotomy repair, nor the difference between them.
  Arms: Music group
Behavioral: Gum Chewing — Women assigned to the gum group will chew plain gum between the beginning and end of the episiotomy repair (15-20 minutes). They will be asked to chew the same brand of easy-to-chew, sugar-free gum that does not contain sorbitol or xylitol. Sugar-free gum is preferred to avoid the risk of GI problems if swallowed with sorbitol-containing gum, and the risk of diarrhea if consumed in excess with xylitol. Given the risk of aspiration while chewing gum, the woman will be positioned in a semi-fowler position.
  Arms: Gum Chewing group

SUMMARY:
Lacerations and episiotomies are serious procedures requiring surgical stitches. Therefore, pain occurs during episiotomy repair. Pain during episiotomy repair also causes anxiety, which in turn exacerbates pain. The goal of pain management is to alleviate pain without experiencing side effects. Midwives and nurses responsible for labor management play an active role in the use of nonpharmacological interventions to manage pain and anxiety during episiotomy repair.

No studies in the literature have been found that combine music and chewing gum during episiotomy repair. This study aims to determine the effects of music and chewing gum during episiotomy repair on pain, anxiety, and patient satisfaction.

This study will be to determine the effects of music and chewing gum during episiotomy repair on pain, anxiety, and patient satisfaction.

DETAILED DESCRIPTION:
Midwives and nurses responsible for labor management play an active role in the use of nonpharmacological interventions to manage pain and anxiety during episiotomy repair.

This study will be a three-group randomized controlled trial to determine the effects of music and chewing gum during episiotomy repair on pain, anxiety, and patient satisfaction.

Research Location and Time Research data collection will be conducted in the delivery room at Adana City Training and Research Hospital between December 2025 and February 2026.

2.3. Research Population and Sample The research population will consist of women who underwent vaginal delivery and episiotomy repair in the delivery room at Adana Training and Research Hospital who meet the study criteria. The research sample will be calculated using a power analysis following a preliminary study (10 music groups, 10 chewing gum groups, and 10 control groups)

Data Collection Tools Data will be a Pregnancy Information Form, a Labor Monitoring Form, Visual Analog Scale (VAS) Pain Score , the State Anxiety Inventory and the Patient Perception of Nursing Care Scale.

Data Collection: Pregnant women participating in the study will be administered an informed consent form, a Pregnancy Information Form, and a Labor Monitoring Form during the first stage of labor. In our study, the VAS pain score will be administered four times: before the episiotomy, during the internal episiotomy repair (suturing at the hymenal ring level), during the external episiotomy repair, and one hour after the episiotomy.

Research Implementation Process After obtaining written and verbal consent from the pregnant women, they will be assigned to the previously determined groups through randomization.

Randomization The name of each group (Music Group, Chewing Gum Group, and Control Group) will be written on a piece of paper, and the group numbers (1, 2, and 3) will be determined by lottery. To ensure randomization in the study, a random number table will be created by entering the number of samples (sample numbers 1, 2, 3, 4, 5, etc.) on the site www.random.org/ and dividing the participants into three groups.

Intervention Group Implementation Steps The music and chewing gum application and other data forms will be introduced to the pregnant women at the beginning of the active phase. Pregnant women participating in the study will be asked to choose relaxing music from an international platform that utilizes the sounds of relaxing music therapies.

Music group protocol: Women in the music group will listen to their preferred music using an connected to speakers in the delivery room between the beginning and end of the episiotomy repair (15-20 minutes).

Chewing Gum group protocol: Women assigned to the chewing gum group will chew plain gum between the beginning and end of the episiotomy repair (15-20 minutes).

Control group implementation steps Pregnant women in the control group will be administered an informed consent form, a Pregnancy Information Form, and a Labor Monitoring Form during the active phase of the first stage.

Data Evaluation Data obtained from the study will be analyzed using the Statistical Package for Social Sciences (SPSS 23.0) for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Study participation criteria

  * Women aged 18-49,
  * Primiparous,
  * Having a medio-lateral episiotomy,
  * Having a singleton pregnancy,
  * Vertex presentation,
  * Having given birth vaginally,
  * Having an episiotomy length of 4-5 cm,
  * Having an uncomplicated newborn,
  * Volunteering to participate in the study,
  * Being able to speak and understand Turkish.

Exclusion Criteria:

* Women who experienced deep lacerations (anal sphincter injuries, 3rd and 4th degree lacerations) during labor,
* Those who underwent operative delivery (with vacuum or forceps),
* Those with visual, hearing, or sensory impairments,
* Those who were not diagnosed with a psychiatric disorder but had problems,
* Those diagnosed with a high-risk pregnancy,
* Those who had any signs of infection, such as vaginal redness or swelling,
* Those who developed complications during any stage of labor,
* Women with chronic illnesses (diabetes mellitus, thyroid disease, and hypertension) will not be included in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — POSTPARTUM WOMEN
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | The research period for a participant takes approximately 1 day
  The Visual Analog Scale (VAS) is used to assess pain intensity. The scale can be scored from 0 to 10 To be collected through a survey. The collected data were planned to be analyzed using SPSS with mean and standard deviation.
The PATIENT'S PERCEPTION SCALE | The research period for a participant takes approximately 1 day
  The PATIENT'S PERCEPTION SCALE scale was developed by Dopier et al. It was developed to measure patients' perceptions of nursing care and their satisfaction with it. The five-point Likert-type scale includes 15 statements regarding the quality of nursing care. Thus, The scale can be scored from 15 to 75. The scale can be scored from 20 to 80. The collected data were planned to be analyzed using SPSS with mean and standard deviation.
The State Anxiety Scale | The research period for a participant takes approximately 1 day
  The State Anxiety Scale (SAAS) was developed by Spielberger et al. The State Anxiety Scale has 20 items. It is used to measure anxiety symptoms. The items describing emotions and behaviors in the scale are scored on a 4-point Likert-type scale: "(1) Not at all," "(2) A little," "(3) A lot," and "(4) Completely." The scale can be scored from 20 to 80. The scale can be scored from 20 to 80 The collected data were planned to be analyzed using SPSS with mean and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Seda KARAÇAY YIKAR, DOCTOR, Study Chair — Cukurova University; Evşen NAZİK, professor, Study Chair — Cukurova University; Fikriye I ADIGÜZEL, Doctor, Study Chair — Adana City Training and Research Hospital; Ayşe S AKBAY KISA, research ass, Principal Investigator — Suleyman Demirel University

IPD SHARING:
Plan to Share IPD: No